CLINICAL TRIAL: NCT06084039
Title: Reducing the Carbon Footprint of Operating Rooms Through Education on the Effects of Inhalation Anesthetics on Global Warming
Brief Title: Reducing the Carbon Footprint Through Education on the Effects of Inhalation Anesthetics on Global Warming
Status: Completed | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kim Hee Young, Assistant professor for the fund, Pusan National University Yangsan Hospital
Other Study IDs: 05-2023-067
Record Dates: First submitted 2023-09-30; First posted 2023-10-16 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inhalation anesthetics, such as desflurane, are identified as contributors to global warming, with the European Union planning to ban desflurane in 2026 due to its impact. The World Federation of Societies of Anesthesiologists (WFSA) has published guidelines to reduce air pollution related to inhalation anesthetics. Inhalation anesthetics account for a significant portion of carbon dioxide equivalent (CO2e) emissions in hospitals and surgery. Various anesthetics have different global warming potentials (GWP100), with desflurane having the highest GWP100. Nitrous oxide and isoflurane, although having lower GWP100, can also impact the environment negatively. Studies have shown that educating anesthesia staff about the environmental impact of desflurane and nitrous oxide can lead to significant reductions in their usage, resulting in lower CO2e emissions and cost savings. However, in some regions like Korea, awareness of the environmental impact of inhalation anesthetics is limited. The authors plan to analyze the impact of education on anesthesiologists regarding inhalation anesthetics and assess changes in their usage and CO2e emissions in clinical settings. The goal is to demonstrate that education can positively influence environmental outcomes and reduce economic losses.

DETAILED DESCRIPTION:
Environmental issues are a global concern and a problem that everyone must solve together. Recently, there have been efforts to reduce carbon footprint in the medical field. In the field of anesthesiology, as it became known that inhalation anesthetics have a significant impact on global warming, the European Union officially declared in 2022 to ban the use of the inhalation anesthetic desflurane from 2026. Additionally, the World Federation of Societies of Anesthesiologists (WFSA) published guidelines on the use of inhalation anesthetics to reduce air pollution in 2022.

Inhalation anesthetics are known to account for 0.01-0.1% of the total carbon dioxide equivalent (CO2e) contribution to global warming. This is 5% of hospital CO2e and 50% of surgery-related CO2e. Only 5% of the inhalation anesthetic is metabolized in the patient's body, and the remaining 95% is discharged through the anesthetic gas scavenging system of the anesthesia machine and released into the atmosphere without any additional post-processing. Representative inhalation anesthetics that are currently widely used include nitrous oxide (N2O), sevoflurane, desflurane, and isoflurane. Comparing their global warming potential (global warming potential 100, GWP100; which indicates the degree of greenhouse gas effect compared to CO2 over 100 years), nitrous oxide 298, sevoflurane 130, desflurane 2540, and isoflurane 510. Among these, desflurane shows the highest GWP100 and is presumed to be due to its high minimum alveolar concentration. In addition, nitrous oxide and isoflurane have relatively low global warming potential, but they can destroy ozone and, in particular, nitrous oxide has a half-life of 114 years, so it can stay in the atmosphere for a long time and affect global warming.

Several studies have reported significant reductions in CO2e and medical costs along with a reduction in the use of these two anesthetics after educating anesthesia staff on the use of desflurane and nitrous oxide. In one study, desflurane usage was reduced by 95.63% and CO2e was reduced by 87.88%. In another study, desflurane use was reduced from 8.3% to 0.3%, CO2e was reduced from 1,681 to 10, and medical costs were saved by $200,000 over 3 years. In Korea, sevoflurane and desflurane are the most used, but the impact of inhalation anesthetics on global warming is not well-known to clinicians, and there are no related studies.

After educating anesthesiologists about the impact of inhalation anesthetics on global warming, the investigators analyzed the use of inhalation anesthetics and changes in CO2e before and after education in actual clinical situations to determine whether education alone could reduce their use. In addition, the investigators aim to show that this can have a positive impact on global warming and economic losses.

Education on the effects of inhalation anesthetics on global warming was conducted for every anesthesiologist in our hospital, and only medical records were reviewed retrospectively to confirm if there were any changes in choice of inhalation anesthetic, and fresh gas flow before and after receiving the training. Inevitably, patients for whom general anesthesia was performed by untrained anesthesiologists about the effects of inhalation anesthetics on global warming were excluded from the analysis. This is an observational study because there is no intervention applied to the patient, and patients not included in the study are also administered general anesthesia using the same method.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent surgery under general anesthesia performed for 1 month before and after education on the effects of inhalation anesthetics on global warming

Exclusion Criteria:

* Surgery performed under regional anesthesia
* Surgery performed under total intravenous anesthesia
* When the type of inhalation anesthetic is changed during surgery
* Short surgery within 1 hour
* In case of anesthesia by an anesthesiologist who did not attend the education on the effects of inhalation anesthetics on global warming

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received general anesthesia using inhalation anesthetics
Sampling Method: Non-Probability Sample
Enrollment: 4478 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
Concentration of inhalation anesthetic used to maintain general anesthesia | Total time for general anesthesia, up to 24hours
  It is calculated using the average value of the inhalation anesthetic concentration and fresh gas flow rate during the entire anesthesia time, excluding 15 minutes after the start of general anesthesia and 15 minutes before the end of anesthesia. The formula for calculating the total amount of inhalation anesthetic is as follows.
  Total amount of inhalation anesthetic used (mL)=([(Fresh gas flow rate (L/min)*1000)*(concentration of inhalation anesthetic (vol%))]/ Density (kg/cm3))* duration of anesthesia (hrs)
  * Amount of sevoflurane used per hour (mL)
    * ([((MW (kg/mol)*(FGF (L/min)*1000)*(concentration of sevoflurane (vol%)/100)/24400)/1000]*60)/ Density (kg/cm3)
    * [(200 *(FGF*1000)*(vol%/100)/24400)/1000]*60/ 0.00152
  * Amount of desflurane used per hour (mL)
    * ([((MW (kg/mol)*(FGF (L/min)*1000)*(concentration of desflurane (vol%)/100)/24400)/1000]*60)/ Density (kg/cm3)
    * [(168 *(FGF*1000)*(vol%/100)/24400)/1000]*60/ 0.001465
Fresh gas flow rate used to maintain general anesthesia | Total time for general anesthesia, up to 24hours
  It is calculated using the average value of the inhalation anesthetic concentration and fresh gas flow rate during the entire anesthesia time, excluding 15 minutes after the start of general anesthesia and 15 minutes before the end of anesthesia. The formula for calculating the total amount of inhalation anesthetic is as follows.
  Total amount of inhalation anesthetic used (mL)=([(Fresh gas flow rate (L/min)*1000)*(concentration of inhalation anesthetic (vol%))]/ Density (kg/cm3))* duration of anesthesia (hrs)
  * Amount of sevoflurane used per hour (mL)
    * ([((MW (kg/mol)*(FGF (L/min)*1000)*(concentration of sevoflurane (vol%)/100)/24400)/1000]*60)/ Density (kg/cm3)
    * [(200 *(FGF*1000)*(vol%/100)/24400)/1000]*60/ 0.00152
  * Amount of desflurane used per hour (mL)
    * ([((MW (kg/mol)*(FGF (L/min)*1000)*(concentration of desflurane (vol%)/100)/24400)/1000]*60)/ Density (kg/cm3)
    * [(168 *(FGF*1000)*(vol%/100)/24400)/1000]*60/ 0.001465

SECONDARY OUTCOMES:
CO2e (total carbon dioxide equivalent), driving equivalent (equivalent driving distance, distance traveled by car to generate the same amount of greenhouse gases), and medical costs incurred due to the use of inhalation anesthetics | Total time for general anesthesia, up to 24hours
  Based on data examined from medical records, CO2e (total carbon dioxide equivalent), driving equivalent (equivalent driving distance, distance required to drive to generate the same amount of greenhouse gases), and medical costs incurred due to inhalation anesthetics were calculated by Anesthesia cost calculator (https://jscalc.io/calc/do45BOJVrzXMaEGC). The formulas for calculating CO2e (total carbon dioxide equivalent), and driving equivalent are as follows.
  * CO2e (kg) =130 * 200* ((FGF*1000)*(concentration of inhalation anesthetic /100)/24400/1000)*60* duration of anesthesia
  * driving equivalent (km) = CO2e *3.922

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Kim, MD, PhD, Principal Investigator — Pusan National University
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea